CLINICAL TRIAL: NCT05211063
Title: Effects of CROCUVIS+® on Computer Vision Syndrome, Sleep and Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Collaborators: Pharmactive Biotech Products S.L.U (Industry)
Responsible Party: Principal Investigator, Maria del Mar Seguí Crespo, Senior lecturer, PhD, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PHARMACTIVE-21TPA
Record Dates: First submitted 2021-12-10; First posted 2022-01-27 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Computer Vision Syndrome; Sleep Disorder; Mood Disorders
MeSH Terms: conditions — Sleep Wake Disorders; Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saffron extract (Crocus sativus) (Experimental): Daily intake of one tablet for 42 days.
  Interventions: Dietary Supplement: Saffron extract (Crocus sativus)
- Placebo (Placebo Comparator): Daily intake of one tablet for 42 days. This tablet is organoleptically indistinguishable from the experimental tablet.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Saffron extract (Crocus sativus) — Daily intake of one tablet for 42 days.
  Arms: Saffron extract (Crocus sativus)
Dietary Supplement: Placebo — Daily intake of one tablet for 42 days.
  Arms: Placebo

SUMMARY:
Previous research has shown the efficacy of CROCUVIS+® dietary supplement, based on saffron extract, in the proper functioning of visual health, for example, against the development of glaucoma. The main objective of this study is to evaluate the efficacy of CROCUVIS® in computer vision syndrome, sleep and mood disorders in a sample of university students who use digital devices.

ELIGIBILITY:
Inclusion Criteria:

* CVS-Q© score ≥6.
* Age between 18 and 40 years (both inclusive).
* Exposure to digital devices 4 hours a day, at least five days a week or more and maintain the same level of exposure throughout the study period.

Exclusion Criteria:

* Monocular corrected distance visual acuity >0.0 LogMAR.
* Ocular pathology under treatment at the time of the study.
* Previous ocular surgery that could affect the tear film or the ocular surface.
* Ocular Surface Disease Index (OSDI) questionnaire score ≥13.
* Previous diagnosis or history of dry eye syndrome and/or blepharitis.
* Regular (daily) use of rigid or soft contact lenses ≥3 days a week.
* Regular use of any ocular lubricant.
* History of oral intake of dietary supplements, with or without herbal ingredients, intended to contribute, maintain or reduce the risk of suffering diseases related to visual function, mood or sleep within the four weeks before the study enrollment.
* Systemic disease:

  1. Uncontrolled hypertension (systolic/diastolic blood pressure >140/90 mmHg).
  2. Uncontrolled diabetes mellitus (fasting blood glucose level >180 mg/dL).
  3. Rheumatoid arthritis.
  4. Tumor disease.
  5. Active hepatitis (type B and C).
  6. Active infectious disease.
  7. Kidney disease that compromises diuresis.
* Current systemic treatment or in the last 3 months with drugs that may interfere with the results, for example:

  1. Opioids.
  2. Antipsychotics.
  3. Antibiotics (tetracyclines, sulfonamides)
  4. Antiarthritic drugs (hydroxychloroquine)
  5. Hypotensive drugs (beta-blockers)
  6. Anticoagulants (heparin, warfarin, or clopidogrel)
  7. Antidepressants (such as fluoxetine, among others)
  8. Hypnotics (eg, benzodiazepines)
* Habitual smoker and/or alcohol drinker. More than 3 cigarettes per day and/or more than 3 Standard Drink Units (SDU) per week, including weekends. SDU is defined as the consumption of 10 ml of alcohol.
* Regular job with rotating shifts including night shift in the last month (including weekends).
* Pregnancy or breastfeeding (also excludes recent pregnancy within the last 3 months) and women planning to become pregnant.
* Participation in another clinical trial in the last 3 months.
* Take any type of dietary supplements with botanical components in the last month.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline computer vision syndrome at 14, 28 and 42 days | 0 (baseline), 14, 28 and 42 days
  Measured with the Computer Vision Syndrome Questionnaire (CVS-Q©). It evaluates the frequency and intensity with which 16 symptoms are perceived over the time of use of digital devices. The score ranges from 0 to 32; computer vision syndrome is considered ≥6. The higher score a subject gained, the worsen ocular condition he/she experienced.
Change from baseline sleep disorders at 14, 28 and 42 days | 0 (baseline), 14, 28 and 42 days
  Measured with the Insomnia Severity Index (ISI). It evaluates 7 items. The score ranges from 0 to 28 (worst). Each item is evaluated on a 5-point Likert scale (from 0 to 4). The final score is obtained from the sum of the responses of all items; insomnia is considered ≥8.
Change from baseline mood at 14, 28 and 42 days | 0 (baseline), 14, 28 and 42 days
  Measured with the Profile of Mood States (POMS). It evaluates 58 items that form 6 factors (tension, depression, anger, vigour, fatigue, and confusion). The score ranges from 68 to 300 (worst mood). Each item is evaluated with a 5-point Likert scale (from 0 to 4). The score of each factor is obtained from the sum of the responses of all the items that define it.
  Total Mood Disturbance = 100+ (Tension + Depression + Anger + Fatigue + Confusion) - Vigour

SECONDARY OUTCOMES:
Change from baseline quality of life related to health at 42 days | 0 (baseline) and 42 days
  Measured with Short Form-36 survey (SF-36). It evaluates 36 items that form 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, mental health). The scores are weighted sums of the questions in each section. The score ranges from 0 to 100. Lower scores = more disability, higher scores = less disability.
Satisfaction question | Last visit (42 day)
  A single satisfaction question. Participants must respond by selecting a number from a Likert scale from 0 to 5.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alicante, San Vicent del Raspeig, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No